CLINICAL TRIAL: NCT01008436
Title: Blood Sparing Strategies: Omni-stat Routinary Use in Cardiac Surgery. A Prospective Randomized Study.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of product due to industrial changes in the manufacturing process altering the final product.
Sponsor: Cardiochirurgia E.H. (Other)
Responsible Party: Principal Investigator, Luca Weltert, Project Leader Luca Weltert, Cardiochirurgia E.H.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00-03
Record Dates: First submitted 2009-11-03; First posted 2009-11-05 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Hemostasis
Keywords: Ability of topical drug to reduce acute and overall bleeding as well as blood transfusions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Traditional best-practice surgical hemostasis
  Interventions: Drug: Control
- Omni-stat Celox (Experimental): Administration of 6 gr of Omni-stat Celox intraoperatively at the time of Hemostasis
  Interventions: Drug: Omni-stat Celox

INTERVENTIONS:
Drug: Omni-stat Celox — Topical administration of 6 gr of Omnistat Celox
  Arms: Omni-stat Celox
Drug: Control — Traditional surgical Hemostasis
  Arms: Control

SUMMARY:
The study enrolles all consecutive patients undergoing cardiac surgery at the European Hospital, Rome. The population undergoes randomization to receive usual surgical hemostasis or added topical application of Omni-stat Celox.

The two populations are followed up prospectively as regarding blood loss and need for blood transfusions, as well as adverse events at 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing heart surgery

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Number of blood units transfused to the patients after surgery till discharge | 30 days
Percentage of acute bleeding controlled by Hemostasis Tool (surgical technique or Omnistat application) in the defined time frame of 10 minutes | 10 minutes

SECONDARY OUTCOMES:
Blood volume collected in chest drains expressed in milliliters, with partial totals 3, 6 and 12 hours after surgery and final total 24 hours after surgery. | 3, 6, 12, 24 hours
Time needed to achieve Hemostasis using Omnistat as regarding to defined time frames of 1,2,3,5,7,10 minutes | 1,2,3,5,7,10 minutes after application

CONTACTS AND LOCATIONS:
Locations (1):
- European Hospital, Rome, Italy